CLINICAL TRIAL: NCT01652677
Title: Randomized Controlled Single-blind Research "Navigation Repetitive Transcranial Magnetic Stimulation in Stroke Rehabilitation"
Brief Title: Navigation Repetitive Transcranial Magnetic Stimulation in Stroke Rehabilitation
Acronym: NTMSR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Chervyakov Alexander, Researcher, Russian Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMS-001
Record Dates: First submitted 2012-06-28; First posted 2012-07-30 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Stroke
Keywords: navigation transcranial magnetic stimulation; stroke rehabilitation
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low-frequency stimulation (Experimental): Stimulation mode: 1 Hz, 100% MT, 20 minutes, unaffected hemisphere
  Interventions: Procedure: Transcranial magnetic stimulation
- High frequency stimulation (Experimental): Stimulation mode: 10 Hz, 80% MT, 2 seconds - stimulation, 58 seconds - rest. - 8 session; affected hemisphere
  Interventions: Procedure: Transcranial magnetic stimulation
- Sham stimulation (Sham Comparator): Patients will receive standard treatment (kinesotherapy, physiotherapy) and simulate of transcranial magnetic stimulation. Also patients will not know about simulation (blind group)
  Interventions: Procedure: Transcranial magnetic stimulation
- Both hemispheric stimulation (Experimental): Stimulation mode: low-frequency to unaffected hemisphere than high-frequency to affected.
  Interventions: Procedure: Transcranial magnetic stimulation

INTERVENTIONS:
Procedure: Transcranial magnetic stimulation — Transcranial magnetic stimulation is a noninvasive technique for including electrical currents in the cerebral cortex by means of time-varying magnetic fields.
  Other Names: Transcranial magnetic stimulation, brain stimulation

SUMMARY:
The aim of research to study therapeutic possibilities of navigation transcranial magnetic stimulation in stroke rehabilitation, finding optimal protocol.

DETAILED DESCRIPTION:
Stroke is the main cause of long-term disability among adults. Disability following stroke results in significant impairment of patients quality of life. There was a lot of investigations with using Transcranial Magnetic Stimulation (TMS) as effective additional therapy in stroke rehabilitation. In this researches uses different protocols and patient's categories: high-frequency, low-frequency, etc. Using method of navigation transcranial magnetic stimulation with neuroimaging could help in choosing optimal protocol, assess effectiveness of therapy and forming prognosis.

ELIGIBILITY:
Inclusion Criteria:

* a person with confirmed cerebral blood flow by ischemic from 8 days to 3 years in a pool of carotid arteries;
* Persons with acute cerebrovascular accidents related to the severity of stroke scale NIHSS (National Institute of Health Stroke Scale) from 5 to 20 points;
* People with cerebral circulatory assessment on the modified Rankin scale at most 3;
* the availability of informed consent;
* healthy volunteers who gave informed consent to participate in the study.

Exclusion Criteria:

* The presence of an implanted pacemaker, intracardiac catheters, electronic pumps;
* The plight of the patient, requiring the maintenance of vital functions by hardware (mechanical ventilation, continuous application infusomats), including an increase of neurological symptoms after 8 days from the start of CVD, myocardial infarction, venous thrombosis of lower extremities, episodes of pulmonary embolism;
* The severity of neurological deficit, which does not allow the patient to pass on their own 10 meters (you can use additional support);
* Pregnancy or possibility of pregnancy in women of childbearing age (before menopause), according to a pregnancy test;
* The presence of metallic elements or implants in the head region, located closer than 20 cm from the edge of the surface coil magnetic stimulator, with the exception of the mouth (metal brackets, vascular sutures, metal plates that cover the defects of the skull, metallic foreign body in the cranial cavity);
* Identification of epileptiform activity during the screening of EEG before the study;
* Epilepsy or seizures in history;
* Patient refusal to participate in the study;

Exclusion criteria were:

* Identified in the study of the general intolerance of the pulsed magnetic field;
* The development of inclusion in the study after acute myocardial infarction and acute cerebral circulatory disorders;
* Setting the pacemaker, intracardiac catheters, or operations on the brain, requiring the abandonment of metallic objects in the cranial cavity;
* The onset of pregnancy;
* Enhancement of the patient, requiring the maintenance of vital functions by hardware (mechanical ventilation);
* The emergence of an epileptic seizure in response to the rhythmic TMS;
* Patient refusal to continue participation in the study;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Evidence of clinically definite ischemic stroke (focal neurological deficits persisting for more than 24 hours) confirmed by non-investigational CT or MRI | up to 20 days
The emergence of epileptic seizure | up to 20 days

SECONDARY OUTCOMES:
Evaluation of the clinical condition of the patient | up to 20 days
  We plan to use different scales to examine clinical condition of patient: Fugl-Meyer scale, Ashworth scale, Perry scale, test with 10 meters walking, Bartel index, Renkin scale

OTHER OUTCOMES:
Pregnancy | up to 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Ludmila A. Chernikova, Study Chair — Research center of neurology Russian academy of medical science; Michael A Piradov, professor, Principal Investigator — Research center of neurology RAMS
Locations (2):
- Russia (2):
  - Research center of neurology Russian academy of medical science, Moscow
  - Research center of neurology RAMS, Moscow, Volokolamskoe Shosse, 80

REFERENCES:
- [Background] Chernikova LA, Kremneva EI, Cherviakov AV, Saenko IV, Konovalov RN, Piramidov MA, Kozlovskaia IB. [New approaches in the study of neuroplasticity process in patients with central nervous system lesion]. Fiziol Cheloveka. 2013 May-Jun;39(3):54-60. doi: 10.7868/s0131164613030053. Russian. PMID 23885553
- [Result] Mokienko OA, Chervyakov AV, Kulikova SN, Bobrov PD, Chernikova LA, Frolov AA, Piradov MA. Increased motor cortex excitability during motor imagery in brain-computer interface trained subjects. Front Comput Neurosci. 2013 Nov 22;7:168. doi: 10.3389/fncom.2013.00168. eCollection 2013. PMID 24319425